CLINICAL TRIAL: NCT05289401
Title: Analgesic Effect of Ultrasound Guided Errector Spinae Plane Block Versus Ultrasound Guided Caudal Block in Pediatric Open Renal Surgeries: A Randomized Comparative Study.
Brief Title: Analgesic Effect of Ultrasound Guided Errector Spinae Plane Block Versus Ultrasound Guided Caudal Block in Pediatric Open Renal Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Chahenda Salem, M.Sc, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-323-2020
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Analgesia , Open Renal Surgeries
Keywords: erector spinae block , caudal block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB (Active Comparator): Unilateral erector spinae block will be performed in the lateral position . 0.5 mL/Kg of bupivacaine 0.125% will be injected taking care not to exceed the maximum recommended dose (2 mg/kg of bupivacaine)
  Interventions: Other: ultrasound guided blocks
- CB (Active Comparator): caudal block performed in lateral position . bolus of 1.2 ml/Kg bupivacaine 0.125% .
  Interventions: Other: ultrasound guided blocks

INTERVENTIONS:
Other: ultrasound guided blocks — Ultrasound Guided Erector Spinae Plane Block Versus Ultrasound Guided Caudal Block in Pediatric

SUMMARY:
comparison between the erector spinae block and caudal block with the aid of the of ultra sound in children as regard time of request of rescue analgesia , degree of intra and post operative pain relief , effect of hemodynamic stability and incidences of complication in open renal surgeries .

DETAILED DESCRIPTION:
Open Renal surgeries (pyeloplasty and nephrectomy) is associated with significant postoperative pain. Adequate postoperative analgesia is important to allow for early mobilization and discharge of the patients .Systemic opioids are usually not sufficient for pain control after renal surgeries in children. The use of opioid in pediatrics has many side effects such as somnolence, vomiting, and up to respiratory depression.

Neuraxial analgesia is usually required in these operations in combination with general anesthesia. Neuraxial analgesia decreases morbidity, mortality, opiate exposure, shortens post anesthesia recovery room time and hospital stay. However, it is usually associated with many complications as urinary retention and excessive motor block.

Caudal block is the most commonly used neuraxial anesthesia in pediatric patients. It can be used for analgesia in different renal surgeries providing adequate pain relief in the post- operative period .

Paediatric regional anaesthesia (PRA) is one of the most valuable and safe tools to treat perioperative pain and is an essential part of modern anaesthetic practice. It offers many advantages to both the patient and the hospital. It provides excellent pain relief and allows caregivers to use multimodal analgesic techniques and decrease the use of opioids without the complications of neuraxial anesthesia. Considerable progress has been made in the practice of PRA over the past few years including availability of information on safety and incorporation of ultrasound guidance. Novel regional anaesthesia (RA) techniques, especially the anterolateral and the posterolateral trunk blocks, show promise .

The erector spinae plane block (ESPB), one of the posterolateral trunk blocks, was first described by Forero et al. in 2016 and has been used by many anaesthesiologists for perioperative pain relief 4. Its mechanism of action is spreading of local anesthetic into multiple paravertebral spaces after injection into the interfascial space between the transverse process of the vertebrae and the erector spinae muscle. It can be used for postoperative analgesia for longer period and decrease the use of opioids with less complications in several pediatric surgeries including nephrectomy and pyeloplasty.

For this reason, ESPB efficacy will be compared to the caudal block efficacy seeking for a simple, safe and effective regional analgesic technique for renal surgeries in children.

Electrical Cardiometry is a method for the non-invasive determination of stroke volume (SV), cardiac output (CO), stroke volume variation (SVV) and other hemodynamic parameters in adults, children, and neonates and it has been validated against "gold standard" methods such as thermodilution. Several potential mechanisms have been suggested for the action of the ESPB such as paravertebral spread as well as epidural spread of local anesthetic. These mechanisms raise the concern of the possible negative hemodynamic consequences of the ESPB which were not properly investigated .

ELIGIBILITY:
Inclusion Criteria:

* Patients 2-6 years old.
* American society of anesthesiologists classification (ASA) I and II .
* Patients undergoing unilateral open renal surgeries.

Exclusion Criteria:

* Refusal of block.
* Bleeding disorders (platelets count < 150,000; INR >1.5; PC< 60%).
* Skin lesion, wounds or infection at the puncture site.
* Known allergy to local anesthetic drugs.
* Contraindications to neuraxial block as sepsis, severe aortic stenosis, increased intracranial pressure.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
primary outcome | at the time of transfer from PACU and then at 1, 2, 3, 4, 6, 8 and 12 hours postoperatively
  The first time to require rescue analgesia in minutes (from the time of erector spinae block or caudal injection to the first registration of CHEOPS pain score more than 6)

SECONDARY OUTCOMES:
secondary outcome | at time of transfer to PACU and then at 1, 2, 3, 4, 6, 8 and 12 hours.
  Total analgesia consumption in each group in the first 12 hours post-operative period

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, C, Egypt

IPD SHARING:
Plan to Share IPD: Undecided